CLINICAL TRIAL: NCT04941846
Title: The Role of Deep Cerebral Vein Variation in Patients With Angiographic Negative Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020111
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Nimodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: nimodipine and euvolemia — administered nimodipine to prevent vasospasm, and euvolemia was maintained via intravenous hydration

SUMMARY:
The incidence of Rosenthal basilar vein (BVR) variants (deep venous drainage variants) was relatively increased in patients with AN-SAH compared with patients with aneurysms. However, the inclusion criteria for AN-SAH patients in these studies were different. Some studies have investigated both PAN-SAH and NPAN-SAH, while some studies have only investigated PAN-SAH patients. However, we believe that NPAN-SAH may be the bleeding caused by non-BVR variation. Although previous studies did not find any association between NPAN-SAH and BVR variants, the results in their study were different, which may be due to the limited number of cases.

ELIGIBILITY:
Inclusion Criteria:

Patients with negative subarachnoid hemorrhage diagnosed by DSA

Exclusion Criteria:

1. In patients with aneurysms, external ventricular drainage (EVD) alone or decompression craniotomy alone or conservative treatment was performed
2. Have a history of trauma or prior brain injury (stroke, cerebral hemorrhage, etc., with associated chronic changes on CT)
3. Patients with loss of imaging data and severe comorditions prior to onset of SAH

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This project plans to include 296 patients who meet the admission and discharge criteria
Sampling Method: Non-Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
favorable or poor outcome | 1 year
  poor outcome (mRS 2-6) or favorable outcome (mRS 0-1).

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjian Fang, MD, Principal Investigator — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2ndAffiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No